CLINICAL TRIAL: NCT03185403
Title: Comparison of the Hemodynamic Effect Between the Paravertebral Block and Thoracic Epidural in Esophageal Surgery With Thoracotomy .
Brief Title: The Hemodynamic Effect Between Two Types of Anesthesia in Esophageal Surgery
Acronym: HEMOBLOC
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Lille (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: 2012_47; 2013-002317-36 (EudraCT Number)
Record Dates: First submitted 2017-05-30; First posted 2017-06-14 (Actual); Last update posted 2017-06-14 (Actual); Status verified 2017-06

CONDITIONS: Epidural Block; Oesophageal Cancer; Oesophagectomy
Keywords: hemodynamic effect; para vertebral block
MeSH Terms: conditions — Esophageal Neoplasms | interventions — Ropivacaine; Sufentanil

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- continous paravertebral block (Active Comparator): echoguided thoracic continous paravertebral block was placed before the surgery.
  A bolus of 5 ml of ropivacaine 0.2% and 10µg of Sufentanil was injected in the catheter at the end of the abdominal time. A continuous infusion of ropivacaine 0.2% at 4ml/h was then initiated at the thoracic time. Postoperative patient-controlled analgesia consisted on an infusion of ropivacaine 0.2% at 6ml/h and a permitted bolus of 4ml every 15min as required.
  Interventions: Other: paravertebral block; Drug: ropivacaine; Drug: Sufentanil
- continous Thoracic epidural block (Active Comparator): thoracic epidural catheter was inserted before the surgery. A bolus of 5 ml of ropivacaine 0.2% and 10µg of Sufentanil was injected in the catheter at the end of the abdominal time. A continuous infusion of ropivacaine 0.2% at 4ml/h was then initiated at the thoracic time. Postoperative patient-controlled analgesia consisted on an infusion of ropivacaine 0.2% at 6ml/h and a permitted bolus of 4ml every 15min as required.
  Interventions: Other: thoracic epidural block; Drug: ropivacaine; Drug: Sufentanil

INTERVENTIONS:
Other: paravertebral block — in the paravertebral block , the catheter was placed under ultrasound echography , at the right thoracic T4/T5 level
  Arms: continous paravertebral block
Other: thoracic epidural block — in the epidural block the catheter was inserted without echography , at T4/T5 level
  Arms: continous Thoracic epidural block
Drug: ropivacaine
Drug: Sufentanil

SUMMARY:
Continuous Paravertebral block (PVB) was reported to provide less episodes of hypotension than continuous thoracic epidural block (TEB). The maintenance of optimal tissue perfusion is essential for esophageal anastomosis in patients undergoing oesophagectomy. the aim of this study is to compare Hemodynamic effect of continous PVB compared to TEB , in patient undergoing oesophagectomy with laparoscopy and thoracotomy.

ELIGIBILITY:
Inclusion Criteria:

* ASA score 1 to 3
* oesophagectomy : abdominal time with laparoscopy ans thoracic time with thoracotomy

Exclusion Criteria:

* pregnancy
* Uncooperative patient
* patient refusal
* Coagulopathy
* allergy to local anesthetic
* Psychological Disorders
* Failure to install the epidural or paravertebral catheter. The patient will therefore be excluded secondarily but will be able to benefit from an alternative technique for the management of his pain.
* Sepsis
* Skin infection at the puncture site
* Allergy to local anesthetics
* Esophagectomy with cervical surgical time
* Patient with chronic pain EVA> 4 before surgery.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 54 (Actual)
Dates: Start 2013-12 (Actual); Primary Completion 2016-07 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
Frequency of hypotension episodes | during perioperative until first 24 hours post operative
  The frequency of hypotension episodes defined by a mean arterial pressure (MAP) less than 70mmHg or a decrease in MAP greater than 20% when compared with the preoperative value

SECONDARY OUTCOMES:
Total amount per patient and per group of vasopressins amines | during perioperative until first 24 hours post operative
Frequency of use of vasopressor agents | during perioperative until first 24 hours post operative
Volumes of fluid administered | during perioperative until the first 24h hours post operative
total amount of morphine consumption | during first 48 hours post operative
visual analog scale | during first 48 hours post operative, at 3 months and 6 months
  Measure the pain severity
DN2 score | during first 48 hours post operative, at 3 months and 6 months
  evaluation with validated scores for chronic and neuropathic pains
Frequency of surgical complications | during first 48 hours post operative
Frequency of pulmonary complications | during first 48 hours post operative
total amount and frequency of Post-operative anti-emetic consumption | during first 48 hours post operative
Death | up to 28 days postoperative

CONTACTS AND LOCATIONS:
Overall Officials: Gilles Lebuffe, MD, PhD, Principal Investigator — University Hospital, Lille
Locations (1):
- CHRU , Hôpital Claude Huriez, Lille, France

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Davies RG, Myles PS, Graham JM. A comparison of the analgesic efficacy and side-effects of paravertebral vs epidural blockade for thoracotomy--a systematic review and meta-analysis of randomized trials. Br J Anaesth. 2006 Apr;96(4):418-26. doi: 10.1093/bja/ael020. Epub 2006 Feb 13. PMID 16476698